CLINICAL TRIAL: NCT06232603
Title: Assessing Medication Adherence in Patients With Chronic Recurrent Multifocal Osteomyelitis
Brief Title: Medication Adherence Intervention in Chronic Recurrent Multifocal Osteomyelitis (CRMO)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of staffing and funding support
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Yongdong (Dan) Zhao, Associate professor, attending physician, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004426
Record Dates: First submitted 2023-10-23; First posted 2024-01-31 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Recurrent Multifocal Osteomyelitis
MeSH Terms: conditions — Chronic recurrent multifocal osteomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education at baseline (Active Comparator): video and ambulatory visit summary (AVS) education will be provided at baseline visit
  Interventions: Other: Education of medication management
- Education at the first follow up (Other): video and AVS education will be provided at the first follow up visit
  Interventions: Other: Education of medication management

INTERVENTIONS:
Other: Education of medication management — Video and handout materials will be provided

SUMMARY:
This project aims to quantify and evaluate rates of non-adherence and barriers to medication adherence in pediatric patients with CRMO followed at Seattle Children's Hospital's robust CRMO program, which is the only clinical program in the Washington, Wyoming, Alaska, Montana, Idaho (WWAMI) region. This will be a stepped-wedge cluster-randomized trial, in which participants will be randomly assigned to one of two groups -- one which receives educational materials at the end of their first clinic visit, and the other which receives educational materials at the end of their second clinic visit. All participants will be given baseline surveys at the start of their first clinic visit, as well as follow-up surveys at the start of their second and third clinic visits. These surveys aim to evaluate rates of non-adherence and qualitative barriers to adherence, as well as efficacy of educational interventions in improving adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRMO
* Receives clinical care at Seattle Children's Hospital
* On one or more scheduled prescription medications

Exclusion Criteria:

-

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Medication possession ratio (MPR) | 6 to 9 months
  The MPR is reported as a percentage calculated as: (total prescription days of supply/ (last prescription date - the first prescription date)). For example, if a patient only filled a one-month prescription twice during 6 months, so only had 60 days of medications available during the 6 months, the MPR would be 33%. A MPR of ≥0.8 is generally accepted as good compliance.
  The MPR data will be calculated for T0 and T1. In order to capture adequate data to calculate the MPR, refill data was acquired for 3 months prior to the beginning of the study (MPR T0) and for 3 months after T1 (MPR T1).

SECONDARY OUTCOMES:
Barriers to adherence | 6-9 months
  A survey will be conducted to determine the barriers predefined and any other barriers

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semo-Oz R, Wagner-Weiner L, Edens C, Zic C, One K, Saad N, Tesher M. Adherence to medication by adolescents and young adults with childhood-onset systemic lupus erythematosus. Lupus. 2022 Oct;31(12):1508-1515. doi: 10.1177/09612033221115974. Epub 2022 Aug 7. PMID 35938626
- [Background] Verma T, Rohan J. Examination of Transition Readiness, Medication Adherence, and Resilience in Pediatric Chronic Illness Populations: A Pilot Study. Int J Environ Res Public Health. 2020 Mar 15;17(6):1905. doi: 10.3390/ijerph17061905. PMID 32183424
- [Background] Saag KG, Bhatia S, Mugavero MJ, Singh JA. Taking an Interdisciplinary Approach to Understanding and Improving Medication Adherence. J Gen Intern Med. 2018 Feb;33(2):136-138. doi: 10.1007/s11606-017-4215-7. No abstract available. PMID 29204970
- [Background] Len CA, Miotto e Silva VB, Terreri MT. Importance of adherence in the outcome of juvenile idiopathic arthritis. Curr Rheumatol Rep. 2014 Apr;16(4):410. doi: 10.1007/s11926-014-0410-2. PMID 24504596
- [Background] Favier LA, Taylor J, Loiselle Rich K, Jones KB, Vora SS, Harris JG, Gottlieb BS, Robbins L, Lai JT, Lee T, Kohlheim M, Gill J, Bouslaugh L, Young A, Griffin N, Morgan EM, Modi AC. Barriers to Adherence in Juvenile Idiopathic Arthritis: A Multicenter Collaborative Experience and Preliminary Results. J Rheumatol. 2018 May;45(5):690-696. doi: 10.3899/jrheum.171087. Epub 2018 Feb 1. PMID 29419467